CLINICAL TRIAL: NCT03970798
Title: A Drug Interaction Study of KW-6356 With Midazolam, Caffeine, or Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6356-005
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Midazolam; Caffeine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KW-6356/Healthy Japanese adult male subjects (Experimental): Period 1: intake of the index substrates at Day 1 (Cohort 1: midazolam, Cohort 2: caffeine + rosuvastatin) followed by Period 2: intake of KW-6356 at Day 4-13, intake of the index substrates at Day 11
  Interventions: Drug: Midazolam; Drug: Caffeine; Drug: Rosuvastatin; Drug: KW-6356

INTERVENTIONS:
Drug: Midazolam — In Period 1, Day 1 a single dose will be administered after fasting for at least 10 hours. In Period 2, Day 11 a single dose will be administered after fasting for at least 10 hours.
Drug: Caffeine — In Period 1, Day 1 a single dose will be administered after fasting for at least 10 hours. In Period 2, Day 11 a single dose will be administered after fasting for at least 10 hours.
Drug: Rosuvastatin — In Period 1, Day 1 a single dose will be administered after fasting for at least 10 hours. In Period 2, Day 11 a single dose will be administered after fasting for at least 10 hours.
Drug: KW-6356 — In Period 2, Day 4-13(except Day11) a single dose of KW-6356 will be administered after breakfast, Day 11 a single dose of KW-6356 will be administered after fasting for at least 10 hours.

SUMMARY:
The purpose of this study is to evaluate the influence of repeated oral doses of KW-6356 on the pharmacokinetics of index substrates for CYP3A4/5, CYP1A2 and BCRP.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals having issued written consent to this study at their own discretion
2. Japanese males aged 20 to 44 years at the time of informed consent
3. Body mass index (BMI) of 18.5 to <25.0 at screening
4. Resting pulse rate of 40 to 100 bpm, systolic blood pressure of 90 to 139 mmHg, and diastolic blood pressure of 40 to 89 mmHg when measured in the supine position at screening

Exclusion Criteria:

1. Individuals with any current disease requiring treatment
2. Individuals having drug allergy or its history
3. Individuals having psychiatric disease or its history
4. Positive results for any of the following infection-related items examined at screening: hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, human T-lymphotropic virus (HTLV)-1 antibody, rapid plasma reagin (PRP) test, Treponema pallidum (TP) antibody.
5. Individuals with clinically significant abnormality detected on 12-lead electrocardiogram (ECG) recorded prior to the first dose of index substrate.
6. Individuals categorized as patients listed in the warnings or contraindications section of the package insert of any of the relevant index substrates (see separate protocol annex 6-8)
7. Individuals having used any drug (including over-the-counter [OTC] drugs, topical agents, vitamin preparations, health supplements, and Chinese herbal medicines) within 2 weeks prior to the first dose of index substrate.
8. Individuals having consumed grapefruit (including any food or beverage containing grapefruit) or any food or beverage containing St John's wort within 1 week prior to the first dose of index substrate.
9. Individuals having smoked or used smoking cessation agents (including chewing or eating of nicotine-containing products and application of nicotine patches) within 4 weeks prior to the first dose of index substrate.
10. Individuals having received inpatient treatment or surgery within 12 weeks prior to the first dose of index substrate.
11. Individuals having participated in a clinical study of a pharmaceutical product or a medical device or any equivalent study and used the investigational product or the unapproved medical device within 16 weeks prior to the first dose of index substrate.
12. Individuals having undergone collection of ≥400 mL of blood within 12 weeks prior to the first dose of index substrate or ≥200 mL of blood within 4 weeks prior to the first dose of index substrate (for blood donation or clinical trial, etc.) or pheresis donation (plateletpheresis or plasmapheresis donation) within 2 weeks prior to the first dose of index substrate.
13. Individuals having issued no consent to adoption of any appropriate contraceptive method during a period from day of admission to 12 weeks after the final dose of the study drug. The appropriate contraceptive method is defined as sexual abstinence or use of 2 of the following contraceptive devices: condom, oral contraceptives, intrauterine device, and pessary.
14. Individuals having received KW-6356 before.
15. Other individuals unsuitable for participating in the study in the opinion of the investigator or subinvestigator.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratio of the major pharmacokinetic parameter (AUC0-t) of the index substrates in combination with or without KW-6356 | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356

SECONDARY OUTCOMES:
Geometric mean ratio of the major pharmacokinetic parameters (Cmax) of the index substrates in combination with or without KW-6356 | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Geometric mean ratio of the major pharmacokinetic parameters (AUC0-∞) of the index substrates in combination with or without KW-6356 | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Pharmacokinetic parameters (tmax) of the index substrates | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Pharmacokinetic parameters (CL/F) of the index substrates | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Pharmacokinetic parameters (Vz/F) of the index substrates | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Pharmacokinetic parameters (t1/2) of the index substrates | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Plasma concentrations of the index substrates | Starting around 2 hours before intake of the index substrates and continued until 24 hours after the last dose of KW-6356
Plasma concentrations of KW-6356 | Starting around 2 hours before intake of KW-6356 and continued until 24 hours after the last dose of KW-6356
Incidence of treatment-emergent adverse events | Starting 24 or 48 hours before intake of the index substrates and continued until 8 days after the last dose of KW-6356

CONTACTS AND LOCATIONS:
Locations (1):
- Fukuoka Mirai Hospital Clinical Research Center, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided